CLINICAL TRIAL: NCT06563414
Title: A Natural History Study of Corneal Abrasions in Patients With Dystrophic Epidermolysis Bullosa (DEB)
Status: Recruiting | Type: Observational
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NHS
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa Dystrophica, Recessive; Epidermolysis Bullosa Dystrophica Dominans
Keywords: Dystrophic Epidermolysis Bullosa; DEB; Corneal Abrasions
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Corneal Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a non-interventional, observational study that will evaluate the natural history of corneal abrasions in patients with Dystrophic Epidermolysis Bullosa (DEB).

DETAILED DESCRIPTION:
The objective of this study is to characterize the natural history of corneal abrasions in patients with Dystrophic Epidermolysis Bullosa (DEB). Patients will be followed via remote weekly symptom diaries and monthly questionnaires to assess corneal abrasion symptoms, frequency, and duration.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or their respective legal guardian must have read, understood, and signed an Institutional Review Board (IRB) approved Informed Consent/Assent Form and must be able to and willing to follow study procedures and instructions.
2. Age 6 months or older at time of Informed Consent/Assent.
3. Prior genetic diagnosis of DEB due to mutation(s) in the collagen type VII alpha 1 chain (COL7A1) gene.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Dystrophic Epidermolysis Bullosa, aged 6 months or older.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Corneal abrasion frequency | Baseline through up to 1 year
  Frequency of corneal abrasion symptoms

SECONDARY OUTCOMES:
Epidermolysis Bullosa Eye Disease Index Symptom Score | Baseline through up to 1 year
  Symptom score for Epidermolysis Bullosa related eye problems, 0 to 30 (higher score indicates worse symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Krystal Biotech, Pittsburgh, Pennsylvania, United States